CLINICAL TRIAL: NCT03390205
Title: Optical Coherence Tomography Angiography in Vitreo and Chorioretinal Pathologies Under the Influence of Dark and Light Adaptation
Brief Title: OCT Angiography in Vitreo and Chorioretinal Pathologies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CRG UZ Brussel (Other)
Responsible Party: Principal Investigator, Pieter Nelis, PhD Candidate, CRG UZ Brussel
Other Study IDs: 2812201748151
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Optical Coherence Tomography
MeSH Terms: interventions — Adaptation, Ocular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Diagnostic Test: Optical coherence tomography angiography under dark and light adaptation
- Controls
  Interventions: Diagnostic Test: Optical coherence tomography angiography under dark and light adaptation

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography angiography under dark and light adaptation — Optical coherence tomography angiography under dark and light adaptation with pupil dilatation

SUMMARY:
In many diseases of the vitreo and chorioretinal complex, perfusion changes have a diagnostic, prognostic or causative role. The visualisation of perfusion was limited to invasive techniques, which were only to depict vasculature in one plane. Optical coherence tomography is able to visualise and quantify eye perfusion layer-specific and non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* Patient with vitreo and chorioretinal pathology, aged-adapted controls

Exclusion Criteria:

* Minors, concomitant ocular pathologies, pregnancy, contra-indication for tropicamide

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with pathology in vitreo and chorioretinal complex and age matched controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Vessel density | 5 minutes after intervention ends
  Vessel density measurements of macula and optic nerve